CLINICAL TRIAL: NCT02590497
Title: The Correlation Between the Genetic and Neuroimaging Signatures in Newly Diagnosed Glioblastoma
Brief Title: Correlation Between the Genetic and Neuroimaging Signatures in Newly Diagnosed Glioblastoma Patients Before Surgery
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: PI made decision
Sponsor: Ohio State University Comprehensive Cancer Center (Other)
Responsible Party: Principal Investigator, Pierre Giglio, Principal Investigator, Ohio State University Comprehensive Cancer Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: OSU-15019; NCI-2015-00873 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2015-09-20; First posted 2015-10-29 (Estimated); Last update posted 2018-01-31 (Actual); Status verified 2018-01

CONDITIONS: Glioblastoma
MeSH Terms: conditions — Glioblastoma | interventions — Gadolinium; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Diagnostic (MRI, tumor tissue analysis) (Experimental): Patients undergo MRI before and after gadolinium contrast administration, including 3D volumetric T1-weighted sequence, FLAIR sequence, diffusion weighted imaging, and perfusion MRI. Tissue samples are also analyzed for the tumor genetic profile.
  Interventions: Procedure: Diffusion Weighted Imaging; Drug: Gadolinium; Other: Laboratory Biomarker Analysis; Procedure: Magnetic Resonance Imaging; Procedure: Perfusion Magnetic Resonance Imaging

INTERVENTIONS:
Procedure: Diffusion Weighted Imaging — Undergo diffusion weighted MRI
  Other Names: Diffusion Weighted MRI; Diffusion-Weighted Magnetic Resonance Imaging; Diffusion-Weighted MR Imaging; Diffusion-Weighted MRI; DWI; DWI MRI; DWI-MRI; MR Diffusion-Weighted Imaging
Drug: Gadolinium — Undergo gadolinium-enhanced MRI
  Other Names: Gd
Other: Laboratory Biomarker Analysis — Tissue genetic analysis
Procedure: Magnetic Resonance Imaging — Undergo gadolinium-enhanced MRI
  Other Names: Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MRI; MRI Scan; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging
Procedure: Magnetic Resonance Imaging — Undergo 3D volumetric T1-weighted sequence
  Other Names: Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MRI; MRI Scan; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging
Procedure: Magnetic Resonance Imaging — Undergo FLAIR sequence
  Other Names: Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MRI; MRI Scan; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging
Procedure: Perfusion Magnetic Resonance Imaging — Undergo perfusion MRI
  Other Names: magnetic resonance perfusion imaging

SUMMARY:
This pilot clinical trial studies the correlation between the genetics and brain images of patients with newly diagnosed glioblastoma before surgery. The genetic characteristics of a tumor are an important way to predict how well it will respond to treatment. Imaging, using magnetic resonance imaging (MRI), takes detailed pictures of organs inside the body, and may also provide information that helps doctors predict how brain tumors will respond to treatment. If MRI can provide doctors with similar information about the tumor as the tumor's genes, it may be able to be used to predict tumor response in patients whose tumors cannot be reached by surgery or biopsy to get tissue samples.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the correlation between the genetic and neuroimaging signature of glioblastoma.

II. Determine the correlation between the neuroimaging signature of glioblastoma and prognosis.

OUTLINE:

Patients undergo MRI before and after gadolinium contrast administration, including 3-dimensional (3D) volumetric T1-weighted sequence, fluid attenuated inversion recovery (FLAIR) sequence, diffusion weighted imaging, and perfusion MRI. Tissue samples are also analyzed for the tumor genetic profile.

ELIGIBILITY:
Inclusion Criteria:

* Patients who will be undergoing surgery for newly-diagnosed glioblastoma
* Subtotal, gross total or biopsy patients will be eligible
* Confirmation of pathology as glioblastoma

Exclusion Criteria:

* Tissue analysis demonstrating pathology other than glioblastoma
* Patients with a contraindication to having MR imaging (e.g. pacemaker) or contrast MR administration (e.g. hypersensitivity to gadolinium or renal insufficiency above the institutional threshold for administration of contrast); patients with hypersensitivity to MR contrast may be able to participate if it has been established that premedication will mitigate the hypersensitivity reaction

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-03-20 (Actual); Primary Completion 2017-10-26 (Actual); Study Completion 2017-10-26 (Actual)

PRIMARY OUTCOMES:
Correlation between the genetic and neuroimaging signature of glioblastoma and prognosis | Day 1
  The average DK parameter and CBV parameter will be compared between classes 1 and 2 based on the 9-gene expression profile at each site using two sample t-test. Data will be transformed or a nonparametric test will be conducted if necessary. Differences in DK and CBV parameters between the two MR techniques (3T MR in OSU and 1.5 T in MUSC) will be explored in each class of patients.
Diffusional kurtosis (DK) values | Day 1
  The average DK parameter and cerebral blood volume (CBV) parameter will be compared between classes 1 and 2 based on the 9-gene expression profile at each site using two sample t-test. Data will be transformed or a nonparametric test will be conducted if necessary. Differences in DK and CBV parameters between the two MR techniques (3T MR in Ohio State University [OSU] and 1.5 T in Medical University of South Carolina [MUSC]) will be explored in each class of patients.
Genetic tumor profile | Day 1
  The average DK parameter and CBV parameter will be compared between classes 1 and 2 based on the 9-gene expression profile at each site using two sample t-test. Data will be transformed or a nonparametric test will be conducted if necessary.

CONTACTS AND LOCATIONS:
Overall Officials: Pierre Giglio, MD, Principal Investigator — Ohio State University Comprehensive Cancer Center

REFERENCES:
- See also: The Jamesline — http://cancer.osu.edu